CLINICAL TRIAL: NCT06073847
Title: Inrebic® (Fedratinib) Post-Marketing Surveillance in Korean Patients With Myelofibrosis
Brief Title: A Post-Marketing Surveillance Study to Assess the Safety of Fedratinib in Korean Patients With Myelofibrosis
Status: Recruiting | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA054-005
Record Dates: First submitted 2023-10-03; First posted 2023-10-10 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Primary Myelofibrosis; Post-polycythemia Vera Myelofibrosis; Post-essential Thrombocythemia Myelofibrosis
MeSH Terms: conditions — Primary Myelofibrosis | interventions — fedratinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with myelofibrosis receiving fedratinib
  Interventions: Drug: Fedratinib

INTERVENTIONS:
Drug: Fedratinib — According to the approved label

SUMMARY:
The purpose of this study is to assess the real-world safety of fedratinib for the treatment of adult participants with primary myelofibrosis (PMF), post polycythemia vera myelofibrosis (post-PV MF), or post essential thrombocythemia myelofibrosis (post-ET MF) who were previously treated with ruxolitinib. Participants will represent the overall patient population with PMF, post-PV MF or post-ET MF who lost adequate response to and/or are intolerant to ruxolitinib. Inadequate response definitions will follow Ministry of Food and Drug Safety-approved label and reimbursement criteria of the Health Insurance Review & Assessment Service.

ELIGIBILITY:
Inclusion Criteria:

* Participants 19 years of age or older
* Participants who will receive fedratinib according to the approved label
* For the first 2 years after marketing authorization, all participants who have received or are receiving fedratinib will also be registered
* Participants who signed the informed consent form

Exclusion Criteria:

* Participants who have been prescribed fedratinib for an indication not approved in Korea
* Participants who have been prescribed fedratinib at a dose not approved in Korea
* Participants for whom fedratinib is contraindicated as clarified in Korean prescribing information approved by the Ministry of Food and Drug Safety

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with primary myelofibrosis, post-polycythemia vera myelofibrosis, or post-essential thrombocythemia myelofibrosis who were previously treated with ruxolitinib
Sampling Method: Non-Probability Sample
Enrollment: 137 (Estimated)
Dates: Start 2023-06-13 (Actual); Primary Completion 2027-12-20 (Estimated); Study Completion 2027-12-20 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events | Up to 6 months
  The type, frequency, seriousness and severity of adverse events (AEs), and relationship of AEs to Inrebic® (fedratinib)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (3):
- South Korea (3):
  - Bristol-Myers Squibb YH, Seoul
  - Local Institution - 0001, Seoul
  - Novotech Laboratory Korea Co., Ltd., Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html